CLINICAL TRIAL: NCT04886687
Title: ROSSETTI: Registry of Combined vs Single Thrombectomy Techniques
Acronym: ROSSETTI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Collaborators: Germans Trias i Pujol Hospital (Other); Hospital Universitari de Bellvitge (Other); University Hospital of Girona Dr. Josep Trueta (Network); Hospital de Cruces (Other); Hospital Universitario Central de Asturias (Other); Hospital Clinico Universitario de Santiago (Other); Hospital San Carlos, Madrid (Other); Hospital Universitario Reina Sofia de Cordoba (Other Government); Hospital Universitario Insular Gran Canaria (Other); Hospital General Universitario de Alicante (Other); Hospital Universitario La Paz (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Sponsor
Other Study IDs: Rossetti
Record Dates: First submitted 2021-04-22; First posted 2021-05-14 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Thrombectomy; Stroke; Ischemic
Keywords: mechanical thrombectomy; stroke
MeSH Terms: conditions — Stroke; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: mechanical thrombectomy — mechanical thrombectomy

SUMMARY:
The ROSSETTI registry is an ongoing investigator-initiated prospective study recruiting deidentified demographic, clinical presentation, site-adjudicated angiographic, procedural, and outcome data in acute ischemic stroke (AIS) consecutive patients treated with mechanical thrombectomy (MT) across 10 Comprehensive Stroke Centers in Spain. The registry started in June 2019 and therefore incorporates the more recent device technology

DETAILED DESCRIPTION:
The study inclusion criteria are the following: age ≥18 years; confirmed large vessel occlusion (LVO) in the anterior circulation (intracranial internal carotid artery M1, proximal M2 segments, time from last seen well to treatment (TLSWT) <24 hours, baseline National Institutes of Health Stroke Scale (NIHSS) score ≥2, and premorbid modified Rankin Scale (mRS) score ≤2. All participating centers received institutional review board approval from their respective institutions and patients or representatives signed informed consent. The study data are collected prospectively through an online questionnaire. Type of stent-retriever , as long as European Community approved, is at the discretion of the operator.

The primary clinical outcome is the rate of excellent clinical outcome, defined as mRS score 0-1 at 90 days (no or minor symptoms but no functional limitations).[28] The primary technical outcome is the rate of first pass effect (FPE) defined as achieving near-complete/complete revascularization [modified Thrombolysis in Cerebral Infarction (mTICI 2c-3)] after single-device and single-pass approach

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* confirmed large vessel occlusion in the anterior circulation (intracranial internal carotid artery, M1segment of middle cerebral artery, proximal M2 segment of middle cerebral artery
* time from last seen well to treatment (TLSWT) <24 hours,
* baseline National Institutes of Health Stroke Scale (NIHSS) score ≥2,
* premorbid modified Rankin Scale (mRS) score ≤2.

Exclusion Criteria:

* No evidence vessel occlusion.
* Extra and Intracranial occlusion or severe stenosis.
* Low platelets (100 x 10000) or impaired function,
* Contraindication of computed tomography or magnetic resonance
* Allergy to iodinated contrast non treatable medically,
* pregnant or breast feeding patient,
* hemorrhagic stroke on computed tomography or Magnetic Resonance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute ischemic stroke due to large vessel occlusion of the anterior circulation
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome | 3 months after thrombectomy
  modified Rankin Score, 0 to 6, higher scores mean a worse outcome
Technical Outcome | 1 day, revascularization grade will be assessed
  Thrombolysis in Cerebral Infarction Scale, 0 to 3, higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Blasco Andaluz, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No